CLINICAL TRIAL: NCT01413386
Title: A Randomized Clinical Trial Comparing Patency and Safety of the Paclitaxel Eluting Covered Metallic Biliary Stent (Niti-S Mira-Cover II Biliary Stent) to the Common Covered Metallic Biliary Stent.
Brief Title: Efficacy and Safety of the Paclitaxel Eluting Covered Biliary Stent to the Common Covered Metallic Biliary Stent
Acronym: MIRAII
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Delayed subject enrollment
Sponsor: Jong Taek, Lee (Industry)
Responsible Party: Sponsor-Investigator, Jong Taek, Lee, Taewoong Medical Co., Ltd., Taewoong Medical Co., Ltd.
Organization: Taewoong Medical Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MIRA-001
Record Dates: First submitted 2011-08-09; First posted 2011-08-10 (Estimated); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Biliary Stricture; Malignant Neoplasms
Keywords: paclitaxel; drug eluting stent
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paclitaxel Eluting Covered Metal Stent (Experimental)
  Interventions: Device: biliary stent
- Covered Metal Stent (Active Comparator)
  Interventions: Device: biliary stent

INTERVENTIONS:
Device: biliary stent — palliative treatment for malignant patients
  Other Names: Niti-S Mira-Cover II Biliary Stent; Niti-S Biliary Stent_ComVi type

SUMMARY:
Paclitaxel covered metal biliary stent is non-inferior to common covered metal biliary stent in their patency rate and safety at the 6 months after stenting.

DETAILED DESCRIPTION:
Paclitaxel covered metal biliary stent (Niti-S Mira-Cover II Biliary Stent) is non-inferior to common covered metal biliary stent (Niti-S Biliary Stent_ComVi type)in their patency rate and safety at the 6 months after stenting.

ELIGIBILITY:
Inclusion Criteria:

* Patient who submitted a written informed consent for the this trial, and 18 ~ 90 years old
* Patient who have pancreatic cancer and/or biliary cancer with mid or distal CBD invasion
* Patient who is inoperable and/or unresectable cases of malignant pancreatic stenosis
* Patient who is attempting of endoscopic biliary metallic stenting (by ERBD) firstly
* Patient who have life expectancy at least longer than 3 months (Karnofsky score >60%)

Exclusion Criteria:

* Patient who previously had surgical biliary drainage
* Patient who carrying bleeding disorder
* Patient who have combined Hilar and/or intra-hepatic duct cancer
* Patient who is improper to endoscopic treatment

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2011-09; Primary Completion 2013-04-18 (Actual); Study Completion 2013-04-23 (Actual)

PRIMARY OUTCOMES:
Accumulative Patency Rate | 6 months

SECONDARY OUTCOMES:
Accumulative Survival Rate | 6 months
Stent migration rate | 6 months
Possibility of Other Treatment after Obstruction | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dong Ki Lee, Ph.D, Study Chair — Kangnam Severance Hospital; Mung Whan Kim, Ph.D, Principal Investigator — Asan Medical Center; Don Haeng Lee, Ph.D, Principal Investigator — Inha University Hospital
Locations (3):
- South Korea (3):
  - In Ha University Hospital, Incheon, In Chun
  - Kangnam Severance Hospital, Kangnam, Seoul
  - Asan Medical Center, Seoul